CLINICAL TRIAL: NCT04436237
Title: Effect of Lower Limb Exproprioception Training in Virtual Environment on Locomotion Performance in Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, Sang-I Lin, Professor, National Cheng Kung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A-ER-108-183
Record Dates: First submitted 2020-06-12; First posted 2020-06-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Spatial Perception; Stroke; Virtual Reality; Exercise Training; Exproprioception
MeSH Terms: conditions — Orientation, Spatial; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non-visual exproprioception training (Experimental): The training requires the participant to place the foot at a target without visual cues of the foot in virtual environment.
  Interventions: Other: Virtual reality foot placement training
- Visual exproprioception group (Active Comparator): The training requires the participant to place the foot at a target with visual cues of the foot in virtual environment.
  Interventions: Other: Virtual reality foot placement training

INTERVENTIONS:
Other: Virtual reality foot placement training — The training is conducted in sitting and standing, and involves both the affected and unaffected foot placement. In the total immersive virtual environment, a target will be presented and the participants are required to move one foot to the target. The location of the moving foot is not seen by the participant in this training.

SUMMARY:
The purpose of this study is to determine if a virtual reality training of foot placement with or without visual cues about the location of the foot in the environment would improve locomotion-related function in persons in the chronic stage of stroke. Participants were randomly assigned to receive twice per week, for a total of 2 weeks' training with visual cues (control group) or without (experimental group). It was hypothesized that the experimental group would be able to place the foot closer to the target when stepping and have more symmetrical gait. So far, 22 stroke patients completed the experiment. Preliminary results support the hypothesis. This project is still ongoing.

ELIGIBILITY:
Inclusion Criteria:

* first time unilateral stroke and onset over 6 months
* able to independent walking with or without aids over 10 meters
* Mini-Mental State Examination (MMSE) score above 24
* orientation intake, able to identify right and left
* normal or corrected-to-normal vision, able to see the 2 cm diameter circle on the floor while standing

Exclusion Criteria:

* gait nearly normal
* had other neurological and musculoskeletal disease which can affect walking ability
* hemineglect
* use virtual reality device will severely discomfort, such as headaches, blurred vision, vertigo or vomiting

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-08-26 (Actual); Primary Completion 2021-12-10 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
foot placement accuracy (cm) | 2 weeks
  The distance between the foot and the target in various stepping tasks
gait symmetry | 2 weeks
  ratio of the two leg step lengths

SECONDARY OUTCOMES:
exproprioception (cm) | 2 weeks
  the error in placing the unaffected foot at a location previously defined by the affected foot

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided